CLINICAL TRIAL: NCT03444441
Title: Estimation of the Minimal Important Difference and Validation of Finnish Versions of Foot and Ankle Patient-reported Outcome Instruments
Brief Title: Estimation of the Minimal Important Difference and Validation of Foot and Ankle Instruments
Status: Completed | Type: Observational
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Central Finland Hospital District (Other); Seinajoki Central Hospital (Other); Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Jussi Repo, Resident surgeon, Central Finland Hospital District
Other Study IDs: FA2018
Record Dates: First submitted 2018-01-13; First posted 2018-02-23 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Foot Diseases; Ankle Disease
Keywords: Foot; Ankle; Finnish; Validation; FAOS; EFAS; LEFS; FAAM; VAS-FA; MOxFA
MeSH Terms: conditions — Foot Diseases | interventions — Fracture Fixation, Internal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Foot or ankle surgery — Surgery for foot or ankle
  Other Names: correction forefoot; correction midfoot; correction hindfoot; correction ankle; combined correction; procedures for osteoarthritis foot or ankle; procedures for instability ankle; correction flatfoot; correction cavus foot; correction equinus foot; procedures for Diabetic ulcer; procedures for Charcot; procedures for tendinopathy Achilles; procedures for tendinopathy other; osteosynthesis; Other foot or ankle surgery

SUMMARY:
The present study investigates the minimal important change and validity of foot and ankle measures.

DETAILED DESCRIPTION:
Patients who are waiting for foot and ankle surgery are recruited from four large referral centers (Peijas Hospital, Seinäjoki Central Hospital, Central Finland Central Hospital, Oulu University Hospital). Participants fill in foot and ankle-specific, generic and sosiodemographic questionnaires on the day of surgery, 6 months after surgery, and 6 months 2 weeks after surgery. Both pen-and-paper and electronic options for completing the questionnaire set are provided.

The data obtained from the Foot and ankle outcome score (FAOS), European foot and ankle society (EFAS) score, modified Lower extremity functional scale (LEFS), Visual analog scale foot and ankle (VAS-FA), Manchester Oxford foot and ankle (MOxFA) questionnaire, and the Foot and ankle ability measure (FAAM) are analyzed using the Rasch Measurement Theory and several other psychometric approaches to investigate minimal important change, reliability, responsiveness and validity of foot and ankle PRO instruments.

ELIGIBILITY:
Inclusion Criteria:

* Full understanding of Finnish language
* Undergoing foot or ankle surgery
* At least 18 years old

Exclusion Criteria:

* Unbalanced mental disorder such as schizophrenia or depression
* Age under 18
* Does not understand Finnish
* Undergoing operation other than foot or ankle

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study recruits adult patients who are undergoing foot or ankle surgery for various reasons.
Sampling Method: Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Minimal important difference | Baseline, 6 months
  Change from baseline scores at 6 months

SECONDARY OUTCOMES:
Reliability | 6 months, 6.5 months
  Change from 6 months scores at 6.5 months
General health question | Baseline, 6 months
  Change from baseline scores at 6 months
General health question | 6 months, 6.5 months
  Change from baseline scores at 6 months
Global assessment scale | 6 months
  Change from baseline scores at 6 months
Validity | Baseline
  Baseline scores
Validity | 6 months
  6 months scores

CONTACTS AND LOCATIONS:
Locations (4):
- Finland (4):
  - Central Finland Central Hospital, Jyväskylä
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - Peijas Hospital, Vantaa

IPD SHARING:
Plan to Share IPD: Undecided